CLINICAL TRIAL: NCT07312045
Title: The Relationship of HALP Score, Blood-Based Inflammatory Indices, and Salivary MMP-8 Levels With Periodontal Disease and Healing After Non-Surgical Periodontal Therapy
Brief Title: HALP Score, Blood-Based Inflammatory Indices, and Salivary MMP-8 in Periodontal Disease and Healing After Non-Surgical Therapy
Status: Recruiting | Type: Observational
Sponsor: Ömer Faruk Okumuş (Other)
Collaborators: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Sponsor-Investigator, Ömer Faruk Okumuş, Assistant Professor, Erzincan University
Organization: Erzincan University (Other)
Other Study IDs: EBYU-HALP-2025
Record Dates: First submitted 2025-11-27; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Periodontal Diseases; Periodontitis; Gingivitis; Chronic
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Periodontally Healthy Individuals: Participants with no clinical signs of gingival inflammation, probing depth ≤3 mm, no clinical attachment loss, and no radiographic bone loss. These individuals serve as the healthy control group.
  Interventions: Procedure: Non-surgical Periodontal Therapy
- Gingivitis Patients: Participants with visible signs of gingival inflammation and bleeding on probing, but without clinical attachment loss or radiographic bone loss. These individuals will receive standard non-surgical periodontal therapy.
  Interventions: Procedure: Non-surgical Periodontal Therapy
- Stage III/IV Periodontitis Patients: Participants diagnosed with stage III or stage IV periodontitis, characterized by clinical attachment loss, probing depth ≥5 mm, and radiographic bone loss. These individuals will receive standard non-surgical periodontal therapy and will be re-evaluated at 3 months.
  Interventions: Procedure: Non-surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non-surgical Periodontal Therapy — Standard full-mouth supra- and subgingival debridement performed in a single session, followed by oral hygiene instructions.

SUMMARY:
This observational clinical study aims to investigate the relationship between the HALP score (Hemoglobin × Albumin × Lymphocyte / Platelet), several blood-based inflammatory indices (including NLR, PLR, LMR, and SII), and salivary MMP-8 levels in individuals with periodontal health, gingivitis, and stage III/IV periodontitis. The study also evaluates how these biomarkers relate to healing following non-surgical periodontal therapy.

A total of 180 participants aged 18-65 years will be included: 50 healthy individuals, 50 patients with gingivitis, and 80 patients with stage III/IV periodontitis. All participants will undergo periodontal clinical examination and provide blood and saliva samples at baseline. Individuals in the gingivitis and periodontitis groups will receive standard non-surgical periodontal treatment (full-mouth debridement) and will return for a 3-month follow-up visit, where periodontal measurements will be repeated. In the periodontitis group, an additional blood sample will be collected at the 3-month follow-up visit.

The primary objective is to determine whether baseline HALP score, systemic inflammatory indices, and salivary MMP-8 levels differ between participants who show good versus poor healing after treatment. Secondary objective include comparing biomarker levels across periodontal status groups. The findings may contribute to early prediction of treatment response and personalized periodontal care.

DETAILED DESCRIPTION:
Following baseline assessments, participants in the gingivitis and periodontitis groups will receive standard non-surgical periodontal therapy. Periodontal clinical measurements will be repeated at the 3-month follow-up visit in these groups. In accordance with the existing ethics committee approval and following further feasibility assessment, an additional blood sample will be collected at the 3-month follow-up visit exclusively from participants in the periodontitis group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Ability to provide informed consent
* No systemic diseases or conditions affecting periodontal status
* For Healthy Group: Probing depth ≤3 mm, no attachment loss, no radiographic bone loss
* For Gingivitis Group: Gingival inflammation and bleeding on probing without attachment loss or bone loss
* For Periodontitis Group: Stage III or stage IV periodontitis according to 2018 classification
* No periodontal treatment within the past 6 months
* Willingness to attend follow-up visits

Exclusion Criteria:

* Systemic diseases influencing periodontal inflammation (e.g., diabetes, autoimmune disorders)
* Current pregnancy or lactation
* Use of antibiotics, anti-inflammatory medications, or immunosuppressive drugs within the last 3 months
* Smokers or individuals using tobacco products
* History of periodontal surgery in the last 6 months
* Presence of fewer than 20 natural teeth
* Any condition that may interfere with study participation or data reliability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals aged 18-65 years presenting to the periodontology clinic for routine examination or periodontal treatment. Participants will be assigned to healthy, gingivitis, or stage III/IV periodontitis groups based on periodontal diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-11-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Differences in Baseline HALP Score Between Good and Poor Treatment Responders | Baseline (T0) to 3 months after treatment (T2)
  Evaluation of whether baseline HALP score differs between good responders (>2 mm reduction in probing depth at sites ≥5 mm) and poor responders (≤2 mm reduction) following non-surgical periodontal therapy in periodontitis patients.

SECONDARY OUTCOMES:
Differences in Baseline NLR Between Good and Poor Responders | Baseline (T0)
  Comparison of baseline neutrophil-to-lymphocyte ratio between good and poor responders in the periodontitis group.
Differences in Baseline PLR Between Good and Poor Responders | Baseline (T0)
  Comparison of baseline platelet-to-lymphocyte ratio between good and poor responders in the periodontitis group.
Differences in Baseline LMR Between Good and Poor Responders | Baseline (T0)
  Comparison of baseline lymphocyte-to-monocyte ratio between good and poor responders in the periodontitis group.
Differences in Baseline SII Between Good and Poor Responders | Baseline (T0)
  Comparison of baseline systemic immune-inflammation index between good and poor responders in the periodontitis group.
Differences in Baseline Salivary MMP-8 Between Good and Poor Responders | Baseline (T0)
  Comparison of baseline salivary MMP-8 levels between good and poor responders in the periodontitis group.
Baseline HALP Score Differences Across Periodontal Status Groups | Baseline (T0)
  Comparison of HALP score among healthy, gingivitis, and stage III/IV periodontitis groups.
Baseline NLR Differences Across Periodontal Status Groups | Baseline (T0)
  Comparison of neutrophil-to-lymphocyte ratio among the three periodontal groups.
Baseline PLR Differences Across Periodontal Status Groups | Baseline (T0)
  Comparison of platelet-to-lymphocyte ratio among the three periodontal groups.
Baseline LMR Differences Across Periodontal Status Groups | Baseline (T0)
  Comparison of lymphocyte-to-monocyte ratio among the three periodontal groups.
Baseline SII Differences Across Periodontal Status Groups | Baseline (T0)
  Comparison of systemic immune-inflammation index among the three periodontal groups.
Baseline Salivary MMP-8 Differences Across Periodontal Status Groups | Baseline (T0)
  Comparison of salivary MMP-8 among healthy, gingivitis, and periodontitis groups.
Changes in Probing Depth After Non-Surgical Periodontal Therapy | Baseline (T0) to 3 months (T2)
  Mean reduction in probing depth from baseline to 3 months in gingivitis and periodontitis patients.
Change in HALP Score After Non-Surgical Periodontal Therapy in Periodontitis Patients | Baseline (T0) to 3 months (T2)
  Evaluation of the change in HALP score from baseline to 3 months after non-surgical periodontal therapy in patients with stage III/IV periodontitis.
Correlations Between Clinical Periodontal Parameters and Biomarker Levels | Baseline (T0)
  Assessment of correlations between probing depth, bleeding on probing, plaque index, clinical attachment level, and biomarkers including HALP score, NLR, PLR, LMR, SII, and salivary MMP-8.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yıldırım University Faculty of Dentistry, Merkez, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided